CLINICAL TRIAL: NCT04779840
Title: Retrospective Study on the Incidence and Management of Anemia in Oncology
Acronym: RESPIRE
Status: Completed | Type: Observational
Sponsor: Weprom (Other)
Responsible Party: Sponsor
Other Study IDs: WP-2019-06
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Anemia; Cancer
MeSH Terms: conditions — Anemia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- period 2011
  Interventions: Other: anemia assessment
- period 2018
  Interventions: Other: anemia assessment

INTERVENTIONS:
Other: anemia assessment — evaluation of anemia status

SUMMARY:
The incidence of anemia ranges from 20 to 75% depending on the type of cancer. It is often present at diagnosis and increases with specific treatments. It has an impact on overall survival and quality of life. Its origins are multiple (pure iron deficiency or functional, malnutrition, dyserythropoiesis, insufficiency renal, hemolysis, chemotherapy, radiotherapy, targeted therapies).

Transfusion is the most common treatment offered in the management of anemia. The incidence of anemia and its consequences are often underestimated during cancer management.

Recommendations were published in 2012. An inventory of the incidence of anemia before and after the publication of these recommendations are proposed in order to assess their impact on daily practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old,
* Follow-up for cancer justifying hospitalization,
* Presenting anemia defined by a hemoglobin level <11 g / dL,
* Patient not having objected to the collection of his data after oral and written information.

Exclusion Criteria:

* patients with a hemoglobin level ≥ 11 g / dL,
* adult patients under guardianship, curatorship or deprived of liberty,
* pregnancy or breast-feeding in progress at the time of hospitalization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cancer and justifying continuous hospitalization for more than one night regardless of pattern.
  Patient informed and not having expressed opposition to the study.
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of anemia | 2 years
  number of patient with anemia (<11.0 g/dL) upon admission to hospital on the number of patients hospitalized over the period

SECONDARY OUTCOMES:
Assessment of transfusion prescriptions | 2 years
  number of transfusions performed on the number of patients hospitalized over the period
Assessment of erythropoiesis stimulating agents (EPO) prescriptions | 2 years
  number of prescriptions for erythropoiesis stimulating agents (EPO)
Assessment of iron prescriptions | 2 years
  number of prescriptions of iron (oral and intravenous)
Time between last transfusion and date of death | 2 years
  Delay between the date of the last transfusion and the date of patient's death
overall survival | 2 years
  Delay between the enrollment date and the date of patient's death

CONTACTS AND LOCATIONS:
Overall Officials: Katell LE DÛ, MD, Principal Investigator — Centre Jean Bernard/Clinique Victor Hugo - LE MANS
Locations (1):
- Centre Jean Bernard - Clinique Victor Hugo, Le Mans, France

IPD SHARING:
Plan to Share IPD: No